CLINICAL TRIAL: NCT05392790
Title: Progressive Resisted Exercise Program Combined with Aerobic Exercise on Osteoporotic Systemic Lupus Erythmatosus Patients, Randomized Controlled Trial
Brief Title: Progressive Resisted Exercise Plus Aerobic Exercise on Osteoporotic Systemic Lupus Erythmatosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003638
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Progressive Resisted Exercise; Aerobic Exercise; Osteoporosis; systemic Lupus Erythmatosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Osteoporosis | interventions — Calcium; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aerobic exercise plus progressive resisted exercise group (Experimental): Will receive aerobic exercise, progressive resisted exercise in addition to traditional care.
  Interventions: Other: Progressive resisted exercise training; Drug: Calcium and Vit D; Other: Aerobic exercises
- Aerobic exercise group (Experimental): Will receive aerobic exercise plus traditional care.
  Interventions: Drug: Calcium and Vit D; Other: Aerobic exercises
- Progressive resisted exercise group (Experimental): Will receive progressive resisted exercise
  Interventions: Other: Progressive resisted exercise training; Drug: Calcium and Vit D
- Control group (Other): Will receive traditional medical treatment in the form of Calcium, Vit D and Bi phosphnate.
  Interventions: Drug: Calcium and Vit D

INTERVENTIONS:
Other: Progressive resisted exercise training — Progressive resisted exercises will be started with the 8 maximum repetition test (8 RM) performed at progressive intensities. The subject will perform the 8 RM test at the beginning and the end of each cycle over the two-month training period. Each training session lasts sixty minutes and will be performed three times per week on alternate days.
  Other Names: Traditional medical treatment
  Arms: Aerobic exercise plus progressive resisted exercise group; Progressive resisted exercise group
Drug: Calcium and Vit D — Traditional medical treatment in the form of Calcium, Vit D and Bi phosphnate.
  Other Names: Bi phosphnate
Other: Aerobic exercises — Aerobic exercises will be applied at 70 - 80% of their maximum heart rate. Trained health professionals supervised the exercise program. Each exercise session will begin with a 5-10-minute warm-up, will be followed by 20 -30 minutes of aerobic activity, and will be concluded with a 5-10-minute cool-down period.
  Other Names: Traditional medical treatment
  Arms: Aerobic exercise group; Aerobic exercise plus progressive resisted exercise group

SUMMARY:
systemic lupus erythematosus (SLE) is the most common autoimmune disease in women of childbearing age. Promoting physical activity is a major national priority for the general population, including patients with chronic diseases. The aim of this study is to investigate the efficiency of combined effect of progressive resisted exercise with aerobic exercise for bone mineral density, quality of life, muscle strength and physical activity for patients with SLE.

DETAILED DESCRIPTION:
The following factors were found to be significantly related to lower BMD by univariate analysis: Caucasian race, older age at diagnosis, higher age at the time of the first DXA, longer disease duration, higher cumulative corticosteroid dose, lower serum levels of 25(OH)D, higher SLE Damage Index score, and postmenopausal status. In the multivariate analysis only the following factors were significant: Caucasian race, increased number of pregnancies, postmenopausal status, higher SLE Damage Index, and higher cumulative corticosteroid dose.

As the quality of life among patients with SLE not fully associated with SLE disease activity, pharmacologic treatments that are effective for SLE disease activity might not be able to improve quality of life in these patients Therefore, the beneﬁt of nonpharmacological therapies on quality of life has been explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus by the classification criteria ACRa and the 2019 EULARb/ACR Classification Criteria for systemic lupus erythematosus
* Systemic Lupus Erythematosus Disease Activity Index ≥4
* For 30 day prior, stable immunosuppressive therapy with steroid (0-20 mg/day) or other immunosuppressive medication such as hydroxychloroquine, chloroquine, azathioprine, methotrexate, mycophenolate mofetil, cyclosporine, belimumab, rituximab

Exclusion Criteria:

* Those who are pregnant.
* Patients with active lupus nephritis, cardiovascular dysfunction, rhythm and conduction disorders.
* Patients with musculoskeletal disturbances; kidney and pulmonary involvements; peripheral neuropathy and fibromyalgia.
* Use of tobacco; treatment with lipid-lowering, chronotropic or antihypertensive drugs

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Systemic lupus erythmatosus is most common in females.
Enrollment: 80 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 6 months
  It will be measured at the lumbar spine and proximal femur by means of dual-energy x-ray absorptiometry (GE Healthcare or Hologic, USA)
Bone Mineral Density | follow up after 3 months
  It will be measured at the lumbar spine and proximal femur by means of dual-energy x-ray

SECONDARY OUTCOMES:
Quality of life (36-Item Short Form Health Survey) | 6 months
  HRQoL using the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36). The SF-36 is a generic measure of HRQoL that contains 36 items grouped into: physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning, emotional role functioning, and mental health. Scores on each subscale range from 0 to 100, with 0 corresponding to the worst health status and 100 to the best health status.
Quality of life (36-Item Short Form Health Survey) | follow up after 3 months
  HRQoL using the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36). The SF-36 is a generic measure of HRQoL that contains 36 items grouped into: physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning, emotional role functioning, and mental health. Scores on each subscale range from 0 to 100, with 0 corresponding to the worst health status and 100 to the best health status.
Muscle strength assessment | 6 months
  will be measured using the Isometric strength. Isometric strength of two lower extremity muscle groups (knee ﬂexors and extensors) will be sampled using an isokinetic exercise machine, the CYBEX (CYBEX International, Inc., Medway, MA).
Muscle strength assessment | follow up after 3 months
  will be measured using the Isometric strength. Isometric strength of two lower extremity muscle groups (knee ﬂexors and extensors) will be sampled using an isokinetic exercise machine, the CYBEX (CYBEX International, Inc., Medway, MA).
Level of physical activity | 6 months
  Patients will be asked to walk up and down a designated corridor in the medical practice for 2min. They will be told to walk at their usual pace and to turn around at the ends of the corridor without stopping.
Level of physical activity | follow up after 3 months
  Patients will be asked to walk up and down a designated corridor in the medical practice for 2min. They will be told to walk at their usual pace and to turn around at the ends of the corridor without stopping.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M Eladl, PhD, Principal Investigator — Assisstant professor of physical therapy for surgery, Faculty of physical therapy
Locations (1):
- Nesma Morgan Allam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Study protocol